CLINICAL TRIAL: NCT03949439
Title: Pre-frailty Status Increases the Risk of Rehospitalization and Mortality in Patients After Cardiac Surgery Without Complications
Brief Title: Pre-frailty and Rehospitalization in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Mayron Faria de Oliveira, Clinical Professor, Instituto Dante Pazzanese de Cardiologia
Other Study IDs: 2.352.465
Record Dates: First submitted 2019-05-12; First posted 2019-05-14 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Frailty Syndrome; Surgery--Complications; Coronary Artery Disease; Valve Anomalies
Keywords: Frailty; Cardiac Suregry; Adverse Events
MeSH Terms: conditions — Frailty; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Frail: non-frail (frailty score 1~3) according to their CFS. Established diagnosis of cardiovascular disease (myocardial infarction, valve regurgitation or stenosis) determined by previous electrocardiogram and/or Doppler echocardiography, and all had surgical interventions (coronary artery bypass [CAB], valve replacement or valve repair). Patients with prior neurological/muscular disease (previous stroke or muscular dystrophies), cognitive impairment resulting from previous injury, frailty score ≥ 5, non-elective/emergency surgery procedures or incomplete data were excluded.
  Interventions: Procedure: Elective Cardiac Surgery
- Pre-Frail: Pre-frail (frailty score 4) according to their CFS. Established diagnosis of cardiovascular disease (myocardial infarction, valve regurgitation or stenosis) determined by previous electrocardiogram and/or Doppler echocardiography, and all had surgical interventions (coronary artery bypass [CAB], valve replacement or valve repair). Patients with prior neurological/muscular disease (previous stroke or muscular dystrophies), cognitive impairment resulting from previous injury, frailty score ≥ 5, non-elective/emergency surgery procedures or incomplete data were excluded.
  Interventions: Procedure: Elective Cardiac Surgery

INTERVENTIONS:
Procedure: Elective Cardiac Surgery — Surgical interventions (coronary artery bypass [CAB], valve replacement or valve repair).

SUMMARY:
Background: It has been demonstrated that pre-frailty has more adverse outcomes after cardiac surgery, however, data on prognosis and long-term evolution in pre-frailty patients after cardiac surgery without postoperative complications are still scarce. Design: To evaluate the impact of pre-frailty on functional survival in patients after cardiac surgery without complications.

DETAILED DESCRIPTION:
A three-year retrospective study based on a physiotherapy database was conducted, and a sample of 453 patients over 65 years of age was enrolled. All of them had an established diagnosis of cardiovascular disease (myocardial infarction, valve regurgitation or stenosis) determined by previous electrocardiogram and/or Doppler echocardiography, and all had surgical interventions (coronary artery bypass [CAB], valve replacement or valve repair). Patients with prior neurological/muscular disease (previous stroke or muscular dystrophies), cognitive impairment resulting from previous injury, frailty score ≥ 5, non-elective/emergency surgery procedures or incomplete data were excluded.

According to the hospital protocol, frailty was assessed by the Clinical Frailty Score (CFS) 24 hours before the scheduled elective surgery. We assigned patients into two groups based on this score: non-frail (frailty score 1~3) and pre-frail (frailty score 4) according to their CFS.

If patients experienced adverse cardiovascular events-both during surgery or at the ICU- such as stroke, infection, prolonged mechanical ventilation time of more than 24 hrs, ICU stay of more than 48 hrs or in-hospital death, they were excluded. We decided to exclude these patients as our objective was to evaluate patients without any surgical complications as our group recently had demonstrated that pre-frail patients had worse outcomes after cardiac surgery in a short period of time.

All included patients were analysed for 3 years using data from the hospital and physiotherapy database, which included medical appointments every 6 months after hospital discharge and major adverse cardiovascular events (atrial fibrillation, pneumonia, pleural effusion, acute myocardial infarction, heart failure, stroke and death).

This retrospective study was approved by the Institutional Ethics Committee (number 2.352.465).

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of cardiovascular disease (myocardial infarction, valve regurgitation or stenosis) determined by previous electrocardiogram and/or Doppler echocardiography, and all had surgical interventions (coronary artery bypass [CAB], valve replacement or valve repair).

Exclusion Criteria:

* neurological/muscular disease (previous stroke or muscular dystrophies), cognitive impairment resulting from previous injury, frailty score ≥ 5, non-elective/emergency surgery procedures or incomplete data

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: established diagnosis of cardiovascular disease (myocardial infarction, valve regurgitation or stenosis) determined by previous electrocardiogram and/or Doppler echocardiography, and all had surgical interventions (coronary artery bypass [CAB], valve replacement or valve repair).
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Adverse Outcome | 3 years after hospital discharge
  atrial fibrillation, pneumonia, pleural effusion, acute myocardial infarction, heart failure, stroke and death

CONTACTS AND LOCATIONS:
Locations (1):
- Dante Pazzanese Institute of Cardiology, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Submit the paper to a medical journal